CLINICAL TRIAL: NCT00537472
Title: Low Dose Spinal Bupivacaine for Total Knee Arthroplasty and Recovery Room Wait Time
Brief Title: Low Dose Spinal Bupivacaine for Total Knee Replacement and Recovery Room Wait Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Melanie Jaeger, MD, FRCPC, Queens University and Kingston General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6106
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Spinal Anesthesia; Total Knee Arthroplasty
Keywords: Bupivacaine; spinal anesthesia; total knee arthroplasty
MeSH Terms: interventions — Anesthesia, Spinal; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental)
  Interventions: Drug: Low dose bupivicaine in spinal anesthetic
- II (Active Comparator)
  Interventions: Drug: Standard dose bupivacaine in spinal anesthetic

INTERVENTIONS:
Drug: Low dose bupivicaine in spinal anesthetic — Bupivacaine 9 mg intrathecal single shot injection at start of surgery
  Arms: I
Drug: Standard dose bupivacaine in spinal anesthetic — Bupivacaine 13 mg intrathecal single shot injection at start of surgery
  Arms: II

SUMMARY:
This study plans to investigate whether a reduced dose of bupivacaine (a local anesthetic numbing drug) injected into the spinal space for a total knee replacement will result in a shorter time to discharge from the recovery room while maintaining adequate surgical anesthesia.

DETAILED DESCRIPTION:
With the doses of bupivacaine currently being used in spinal anesthetics at our institution, patients' sensory blocks are often much higher than needed to achieve adequate surgical anesthesia. This translates into a prolonged waiting period in the recovery room before the level regresses down to the pre-existing standard for discharge to the ward, as well as the pre-existing level before a post-operative nerve block for extended pain relief can be performed. This prolonged period in the recovery room leads to general delays in operating room usage and thus surgical cancellations. The excessive drug doses currently used also put patients at risk for increasing side effects including low blood pressure, slow heart rates, and nausea and vomiting.

By using a reduced dose of bupivacaine in a spinal anesthetic for a one sided knee replacement, we hope to significantly reduce the recovery room waiting times until the criteria for recovery room discharge or completion of a post-operative nerve block are met, while still providing adequate surgical anesthesia.

Patients will receive either 9 mg (intervention dose) or 13 mg (control dose) of bupivacaine through a spinal injection. Once the patients enter the recovery room after surgery the level of their sensory block will be tested as per usual protocol by the recovery room nurses every 15 minutes until a predefined level has been reached, and the two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective one-sided total knee replacement for osteoarthritis at our institution where spinal anesthesia has been chosen by the patient and the anesthetist

Exclusion Criteria:

* Contraindications to spinal anesthesia (such as increase pressure in brain, bleeding disorder, serious valvular heart disease, serious infection in the blood or on your lower back, certain neurological disorders such as multiple sclerosis, desire for a general anesthetic)
* Allergies to local anesthetics, morphine or fentanyl
* Both knees being done at same surgery
* Revision of a previous knee replacement
* Knee replacement for reasons other than osteoarthritis (such as rheumatoid arthritis)
* Potential for difficult intubation in case of need for general anesthetic
* Patients under 150 cm or over 200 cm
* BMI greater than 40
* Lack of patient consent or patient refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Time from spinal injection of bupivicaine until recovery room discharge criteria met. | Until recovery room discharge post surgery

SECONDARY OUTCOMES:
Need for pharmacologic rescue from inadequate spinal block during the procedure. | Until end of surgery
Time from entrance into recovery room until criteria for a recovery room discharge are met | Until recovery room discharge criteria are met
Time from entrance into recovery room until criteria for a femoral nerve block for post-operative pain control are met | Until criteria are met for post operative nerve block in recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Jaeger, MD, FRCPSC, Principal Investigator — Staff anesthesiologist at Kingston General Hospital; Dale Engen, MD, FRCPSC, Study Director — Staff anesthesiologist at Kingston General Hospital; Devin Sydor, MD, Study Director — Anesthesiology resident at Kingston General Hospital/Queen's University
Locations (1):
- Kingston General Hospital, Kingston, Ontario, Canada